CLINICAL TRIAL: NCT06574113
Title: Validation of Cuffless Blood Pressure Measurements Using the Perin Health Patch
Status: Recruiting | Type: Observational
Sponsor: Perin Health Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: PHD-001-24
Record Dates: First submitted 2024-08-23; First posted 2024-08-27 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Blood Pressure
Keywords: Cuffless blood pressure; Wearable device

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: Perin Health Patch — The Perin Health Patch (PHP)is a multimodal wearable health patch, which combines auscultation, electrocardiography (ECG), pulse oximetry via photoplethysmography (PPG), bioimpedance (BioZ), skin temperature, and motion and tilt sensors. The PHP integrates multiwavelength PPG (MWPPG) with blue, green, red, and IR LEDs, allowing for precise calculation of PTT, PWV, and related unique parameters, that are used for the calculation of cuffless blood pressure.

SUMMARY:
This study aims to validate a proprietary cuffless blood pressure algorithm using measurements from a multi-modal chest-worn medical device, the Perin Health Patch (PHP).

DETAILED DESCRIPTION:
The study will compare the performance of the PHP to an ambulatory blood pressure cuff across 85 subjects for a 10-minute monitoring period, followed by an optional cold pressor test and an additional 10-minute monitoring period. The study aims to confirm that the calibrated measurement from the wearable device meets AAMI performance standards.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older,
* Willing and able to provide informed consent,
* Able to comply with study procedure.

Exclusion Criteria:

* Any member defined under 'Special Population' in the AAMI standards (Pregnant, children, arm circumference > 42 cm),
* Patient with a pacemaker,
* History of reactions to medical adhesives,
* Inability to comply with the study procedure,
* Non-English Speaker.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of male and female adult participants aged 18 years or older who are willing and able to provide informed consent and comply with the study procedures. Participants may be healthy or have comorbidities, so long as participants are members of any 'Special Population' as defined by the AAMI standards, including but not limited to pregnant individuals, children, and those with an arm circumference greater than 42 cm. Due to the nature of the investigational device, individuals with pacemakers or a history of reactions to medical adhesives may not participate.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2024-10-15 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Cuffless blood pressure measurement performance | 3 months
  Calculate the mean error and standard deviation of blood pressure (BP) measurements from the PHP relative to the ambulatory blood pressure cuff and determine compliance of the PHP's performance with AAMI standards and ISO 81060-2.

SECONDARY OUTCOMES:
Demographic performance variance | 3 months
  Determine any variations in performance on certain demographic groups, including subjects who are overweight, subjects with dark skin pigmentation, or subjects with comorbidities.

CONTACTS AND LOCATIONS:
Overall Officials: Ian M McLane, Ph.D., Principal Investigator — Perin Health Devices
Locations (1):
- Perin Health Devices, Woodland Hills, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Access to the data will be restricted to the study team. If any future or secondary analysis is conducted by other investigators, a formal approval process will be undertaken, including the validation of proper training certificates and data use plans. Training, requests, and approvals will be maintained in Perin Health Devices' electronic quality management system (eQMS). PI McLane will be responsible for the oversight of the electronic and physical data.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-06-03): https://cdn.clinicaltrials.gov/large-docs/13/NCT06574113/Prot_SAP_ICF_000.pdf